CLINICAL TRIAL: NCT00070174
Title: Treatment of Newly Diagnosed Childhood Acute Myeloid Leukemia (AML) Using Intensive MRC-Based Therapy and Gemtuzumab Ozogamicin (GMTZ): A COG Pilot Study
Brief Title: Gemtuzumab Ozogamicin in Treating Young Patients With Newly Diagnosed Acute Myeloid Leukemia Undergoing Remission Induction and Intensification Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: AAML03P1; CDR0000330133 (Other: Clinical Trials.gov); COG-AAML03P1 (Other: Children's Oncology Group)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Leukemia
Keywords: untreated childhood acute myeloid leukemia and other myeloid malignancies; childhood acute monocytic leukemia (M5b); childhood acute megakaryocytic leukemia (M7); childhood acute minimally differentiated myeloid leukemia (M0); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myelomonocytic leukemia (M4); childhood acute monoblastic leukemia (M5a); childhood acute erythroleukemia (M6)
MeSH Terms: conditions — Leukemia | interventions — Asparaginase; Busulfan; Cyclophosphamide; Cyclosporine; Cytarabine; Daunorubicin; Etoposide; Gemtuzumab; Methotrexate; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: asparaginase
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: etoposide
Drug: gemtuzumab ozogamicin
Drug: methotrexate
Drug: mitoxantrone hydrochloride
Procedure: allogeneic bone marrow transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor bone marrow transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. Also, monoclonal antibodies, such as gemtuzumab ozogamicin, can find cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying how well gemtuzumab ozogamicin works in treating young patients who are undergoing remission induction, intensification therapy, and allogeneic bone marrow transplant for newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of gemtuzumab ozogamicin in children with newly diagnosed acute myeloid leukemia undergoing intensive remission induction and intensification therapy.
* Determine the complete remission rate of patients treated with this regimen.

Secondary

* Determine the feasibility of performing biological studies (e.g., FLT3-ITD and MRD) for risk group stratification in these patients.
* Determine the effect of karyotypic abnormalities on survival in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Induction I: Patients receive high-dose cytarabine (ARA-C) IV twice daily on days 1-10; daunorubicin IV over 6 hours on days 1, 3, and 5; etoposide IV over 4 hours on days 1-5; and gemtuzumab ozogamicin IV over 2 hours on day 6. Patients with CNS-negative disease receive ARA-C intrathecally (IT) on day 1. Patients with CNS-positive disease receive ARA-C IT twice weekly for 2-3 weeks. Between days 28-35, patients are evaluated. Patients achieving remission or who have no more than 20% blasts proceed to induction II.
* Induction II: Patients receive ARA-C IV twice daily on days 1-8; ARA-C IT on day 1; and daunorubicin IV and etoposide IV as in induction I. Between days 28-35 patients are evaluated. Patients achieving complete remission proceed to intensification course I.
* Intensification course I: Patients receive ARA-C IV over 1 hour twice daily on days 1-5; ARA-C IT as in induction II; and etoposide IV over 1 hour on days 1-5. Patients are evaluated at day 28. Patients with a 5/6 or 6/6 matched family donor proceed to allogeneic bone marrow transplantation. All other patients in complete remission proceed to intensification course II.
* Intensification course II: Patients receive ARA-C IV over 2 hours twice daily on days 1-4; ARA-C IT as in induction II; mitoxantrone IV over 1 hour on days 3-6; and gemtuzumab ozogamicin IV over 2 hours on day 7. Patients are evaluated on day 28 and then proceed to intensification course III.
* Intensification course III: Patients receive ARA-C IV over 3 hours twice daily on days 1, 2, 8, and 9 and asparaginase intramuscularly on days 2 and 9.
* Allogeneic bone marrow transplantation: Patients receive a preparative regimen comprising busulfan IV over 2 hours 4 times daily on days -9 to -6 and cyclophosphamide IV over 1 hour once daily on days -5 to -2. Allogeneic stem cells are infused on day 0.
* Graft-versus-host disease prophylaxis: Patients receive oral or IV cyclosporine twice daily on days -1 to 50 and methotrexate IV once daily on days 1, 3, 6, and 11.

In all courses, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 6 months, every 2 months for 6 months, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 330 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed primary acute myeloid leukemia (AML)

  * At least 20% bone marrow blasts
  * Meets the customary FAB criteria for AML

    * Patients with cytopenias and bone marrow blasts who do not meet the FAB criteria are eligible provided they have a karyotypic abnormality characteristic of de novo AML (e.g., t[8;21], inv16, or t[16;16]) OR they have the unequivocal presence of megakaryoblasts
  * Isolated granulocytic sarcoma (myeloblastoma) allowed regardless of the results outlined above
* Previously untreated disease
* No promyelocytic leukemia (FAB M3)
* No documented myelodysplastic syndromes (preleukemia) (e.g., chronic myelomonocytic leukemia, refractory anemia [RA], RA with excess blasts, or RA with ringed sideroblasts)
* No juvenile myelomonocytic leukemia
* No Fanconi's anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndrome
* No Down syndrome

PATIENT CHARACTERISTICS:

Age

* 1 month to 21 years* NOTE: *Children under 1 month of age who have progressive disease are allowed

Performance status

* Karnofsky 50-100% (over 16 years of age) OR
* Lansky 50-100% (ages 1 to 16)* NOTE: Children under 1 year of age do not require a performance status

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No inadequate liver function

Renal

* No inadequate renal function
* No hyperuricemia (greater than 8.0 mg/dL)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) at least 70 mL/min OR an equivalent normal GFR OR
* Creatinine no greater than 1.5 times normal

Cardiovascular

* Shortening fraction at least 27% by echocardiogram OR
* Ejection fraction at least 50% by MUGA

Pulmonary

* No proven or suspected pneumonia

Other

* Not pregnant or nursing
* No proven or suspected sepsis or meningitis

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy except intrathecal cytarabine administered that was administered at diagnosis

Endocrine therapy

* Prior topical and inhalation steroids allowed
* No concurrent steroids as antiemetics

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Other

* No prior antileukemic therapy
* No concurrent pressor agent or ventilatory support unless approved by the study chair
* No concurrent participation in another COG therapeutic study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2003-12; Primary Completion 2006-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety
Complete remission rate

SECONDARY OUTCOMES:
Feasibility
Effect of karyotypic abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Janet Franklin, MD, MPH, Study Chair — Children's Hospital Los Angeles
Locations (148):
- United States (134):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center - Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Hartford, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, East Lansing, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Point Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Children's Hospitals and Clinics - Minneapolis/St. Paul, Minneapolis, Minnesota
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Brooklyn Hospital Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Office of S. David Lang, Herston, Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (9):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Swiss Pediatric Oncology Group Bern, Bern, Chihuahua, Switzerland

REFERENCES:
- [Background] Pollard JA, Alonzo TA, Loken M, Gerbing RB, Ho PA, Bernstein ID, Raimondi SC, Hirsch B, Franklin J, Walter RB, Gamis A, Meshinchi S. Correlation of CD33 expression level with disease characteristics and response to gemtuzumab ozogamicin containing chemotherapy in childhood AML. Blood. 2012 Apr 19;119(16):3705-11. doi: 10.1182/blood-2011-12-398370. Epub 2012 Feb 29. PMID 22378848
- [Background] Ho PA, Kopecky KJ, Alonzo TA, Gerbing RB, Miller KL, Kuhn J, Zeng R, Ries RE, Raimondi SC, Hirsch BA, Oehler V, Hurwitz CA, Franklin JL, Gamis AS, Petersdorf SH, Anderson JE, Godwin JE, Reaman GH, Willman CL, Bernstein ID, Radich JP, Appelbaum FR, Stirewalt DL, Meshinchi S. Prognostic implications of the IDH1 synonymous SNP rs11554137 in pediatric and adult AML: a report from the Children's Oncology Group and SWOG. Blood. 2011 Oct 27;118(17):4561-6. doi: 10.1182/blood-2011-04-348888. Epub 2011 Aug 26. PMID 21873548
- [Background] Ho PA, Kuhn J, Gerbing RB, Pollard JA, Zeng R, Miller KL, Heerema NA, Raimondi SC, Hirsch BA, Franklin JL, Lange B, Gamis AS, Alonzo TA, Meshinchi S. WT1 synonymous single nucleotide polymorphism rs16754 correlates with higher mRNA expression and predicts significantly improved outcome in favorable-risk pediatric acute myeloid leukemia: a report from the children's oncology group. J Clin Oncol. 2011 Feb 20;29(6):704-11. doi: 10.1200/JCO.2010.31.9327. Epub 2010 Dec 28. PMID 21189390
- [Background] Ho PA, Alonzo TA, Kopecky KJ, Miller KL, Kuhn J, Zeng R, Gerbing RB, Raimondi SC, Hirsch BA, Oehler V, Hurwitz CA, Franklin JL, Gamis AS, Petersdorf SH, Anderson JE, Reaman GH, Baker LH, Willman CL, Bernstein ID, Radich JP, Appelbaum FR, Stirewalt DL, Meshinchi S. Molecular alterations of the IDH1 gene in AML: a Children's Oncology Group and Southwest Oncology Group study. Leukemia. 2010 May;24(5):909-13. doi: 10.1038/leu.2010.56. Epub 2010 Apr 8. PMID 20376086
- [Background] Ho PA, Zeng R, Alonzo TA, Gerbing RB, Miller KL, Pollard JA, Stirewalt DL, Heerema NA, Raimondi SC, Hirsch B, Franklin JL, Lange B, Meshinchi S. Prevalence and prognostic implications of WT1 mutations in pediatric acute myeloid leukemia (AML): a report from the Children's Oncology Group. Blood. 2010 Aug 5;116(5):702-10. doi: 10.1182/blood-2010-02-268953. Epub 2010 Apr 22. PMID 20413658
- [Background] Phillips CL, Gerbing R, Alonzo T, Perentesis JP, Harley IT, Meshinchi S, Bhatla D, Radloff G, Davies SM. MDM2 polymorphism increases susceptibility to childhood acute myeloid leukemia: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2010 Aug;55(2):248-53. doi: 10.1002/pbc.22519. PMID 20582981
- [Background] Pollard JA, Alonzo TA, Gerbing RB, Ho PA, Zeng R, Ravindranath Y, Dahl G, Lacayo NJ, Becton D, Chang M, Weinstein HJ, Hirsch B, Raimondi SC, Heerema NA, Woods WG, Lange BJ, Hurwitz C, Arceci RJ, Radich JP, Bernstein ID, Heinrich MC, Meshinchi S. Prevalence and prognostic significance of KIT mutations in pediatric patients with core binding factor AML enrolled on serial pediatric cooperative trials for de novo AML. Blood. 2010 Mar 25;115(12):2372-9. doi: 10.1182/blood-2009-09-241075. Epub 2010 Jan 7. PMID 20056794
- [Background] Berman JN, Gerbing RB, Alonzo TA, Ho PA, Miller K, Hurwitz C, Heerema NA, Hirsch B, Raimondi SC, Lange B, Franklin JL, Gamis A, Meshinchi S. Prevalence and clinical implications of NRAS mutations in childhood AML: a report from the Children's Oncology Group. Leukemia. 2011 Jun;25(6):1039-42. doi: 10.1038/leu.2011.31. Epub 2011 Mar 1. No abstract available. PMID 21358716
- [Background] Ho PA, Alonzo TA, Gerbing RB, Pollard J, Stirewalt DL, Hurwitz C, Heerema NA, Hirsch B, Raimondi SC, Lange B, Franklin JL, Radich JP, Meshinchi S. Prevalence and prognostic implications of CEBPA mutations in pediatric acute myeloid leukemia (AML): a report from the Children's Oncology Group. Blood. 2009 Jun 25;113(26):6558-66. doi: 10.1182/blood-2008-10-184747. Epub 2009 Mar 20. PMID 19304957
- [Background] Sung L, Alonzo TA, Gerbing RB, Aplenc R, Lange BJ, Woods WG, Feusner J, Franklin J, Patterson MJ, Gamis AS; Children's Oncology Group. Respiratory syncytial virus infections in children with acute myeloid leukemia: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2008 Dec;51(6):784-6. doi: 10.1002/pbc.21710. PMID 18680152
- [Background] Pollard J, Alonzo T, Gerbing R, et al.: Prevalence and prognostic significance of c-KIT mutations in pediatric CBF AML patients enrolled on serial CCG/COG protocols. [Abstract] Blood 110 (11): A-1442, 2007.
- [Result] Cooper TM, Franklin J, Gerbing RB, Alonzo TA, Hurwitz C, Raimondi SC, Hirsch B, Smith FO, Mathew P, Arceci RJ, Feusner J, Iannone R, Lavey RS, Meshinchi S, Gamis A. AAML03P1, a pilot study of the safety of gemtuzumab ozogamicin in combination with chemotherapy for newly diagnosed childhood acute myeloid leukemia: a report from the Children's Oncology Group. Cancer. 2012 Feb 1;118(3):761-9. doi: 10.1002/cncr.26190. Epub 2011 Jul 15. PMID 21766293
- [Result] Gudgeon CJ, Harrington KH, Laszlo GS, Alonzo TA, Gerbing RB, Gamis AS, Raimondi SC, Hirsch BA, Meshinchi S, Walter RB. High expression of neutrophil elastase predicts improved survival in pediatric acute myeloid leukemia: a report from the Children's Oncology Group. Leuk Lymphoma. 2013 Jan;54(1):202-4. doi: 10.3109/10428194.2012.700480. Epub 2012 Jul 9. No abstract available. PMID 22680764
- [Result] Loken MR, Alonzo TA, Pardo L, Gerbing RB, Raimondi SC, Hirsch BA, Ho PA, Franklin J, Cooper TM, Gamis AS, Meshinchi S. Residual disease detected by multidimensional flow cytometry signifies high relapse risk in patients with de novo acute myeloid leukemia: a report from Children's Oncology Group. Blood. 2012 Aug 23;120(8):1581-8. doi: 10.1182/blood-2012-02-408336. Epub 2012 May 30. PMID 22649108
- [Result] Ho PA, Kutny MA, Alonzo TA, Gerbing RB, Joaquin J, Raimondi SC, Gamis AS, Meshinchi S. Leukemic mutations in the methylation-associated genes DNMT3A and IDH2 are rare events in pediatric AML: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2011 Aug;57(2):204-9. doi: 10.1002/pbc.23179. Epub 2011 Apr 18. PMID 21504050
- [Result] Walter RB, Alonzo TA, Gerbing RB, Ho PA, Smith FO, Raimondi SC, Hirsch BA, Gamis AS, Franklin JL, Hurwitz CA, Loken MR, Meshinchi S. High expression of the very late antigen-4 integrin independently predicts reduced risk of relapse and improved outcome in pediatric acute myeloid leukemia: a report from the children's oncology group. J Clin Oncol. 2010 Jun 10;28(17):2831-8. doi: 10.1200/JCO.2009.27.5693. Epub 2010 Apr 26. PMID 20421533
- [Result] Walter RB, Alonzo TA, Gerbing RB, et al.: High expression of the very late antigen (VLA)-4 (CD49d) integrin predicts for reduced risk of relapse and better outcome in pediatric acute myeloid leukemia (AML): A report from the Children's Oncology Group. [Abstract] Blood 114 (22): A-1592, 2009.
- [Result] Franklin J, Alonzo T, Hurwitz CA, et al.: COG AAML03P1: efficacy and safety in a pilot study of intensive chemotherapy including gemtuzumab in children newly diagnosed with acute myeloid leukemia (AML). [Abstract] Blood 112 (11): A- 136, 2008.
- [Derived] Tarlock K, Gerbing RB, Ries RE, Smith JL, Leonti A, Huang BJ, Kirkey D, Robinson L, Peplinski JH, Lange B, Cooper TM, Gamis AS, Kolb EA, Aplenc R, Pollard JA, Alonzo TA, Meshinchi S. Prognostic impact of cooccurring mutations in FLT3-ITD pediatric acute myeloid leukemia. Blood Adv. 2024 May 14;8(9):2094-2103. doi: 10.1182/bloodadvances.2023011980. PMID 38295280
- [Derived] Zarnegar-Lumley S, Alonzo TA, Gerbing RB, Othus M, Sun Z, Ries RE, Wang J, Leonti A, Kutny MA, Ostronoff F, Radich JP, Appelbaum FR, Pogosova-Agadjanyan EL, O'Dwyer K, Tallman MS, Litzow M, Atallah E, Cooper TM, Aplenc RA, Abdel-Wahab O, Gamis AS, Luger S, Erba H, Levine R, Kolb EA, Stirewalt DL, Meshinchi S, Tarlock K. Characteristics and prognostic impact of IDH mutations in AML: a COG, SWOG, and ECOG analysis. Blood Adv. 2023 Oct 10;7(19):5941-5953. doi: 10.1182/bloodadvances.2022008282. PMID 37267439
- [Derived] Bertrums EJM, Smith JL, Harmon L, Ries RE, Wang YJ, Alonzo TA, Menssen AJ, Chisholm KM, Leonti AR, Tarlock K, Ostronoff F, Pogosova-Agadjanyan EL, Kaspers GJL, Hasle H, Dworzak M, Walter C, Muhlegger N, Morerio C, Pardo L, Hirsch B, Raimondi S, Cooper TM, Aplenc R, Gamis AS, Kolb EA, Farrar JE, Stirewalt D, Ma X, Shaw TI, Furlan SN, Brodersen LE, Loken MR, Van den Heuvel-Eibrink MM, Zwaan CM, Triche TJ, Goemans BF, Meshinchi S. Comprehensive molecular and clinical characterization of NUP98 fusions in pediatric acute myeloid leukemia. Haematologica. 2023 Aug 1;108(8):2044-2058. doi: 10.3324/haematol.2022.281653. PMID 36815378
- [Derived] Vujkovic M, Attiyeh EF, Ries RE, Goodman EK, Ding Y, Kavcic M, Alonzo TA, Wang YC, Gerbing RB, Sung L, Hirsch B, Raimondi S, Gamis AS, Meshinchi S, Aplenc R. Genomic architecture and treatment outcome in pediatric acute myeloid leukemia: a Children's Oncology Group report. Blood. 2017 Jun 8;129(23):3051-3058. doi: 10.1182/blood-2017-03-772384. Epub 2017 Apr 14. PMID 28411282